CLINICAL TRIAL: NCT03774082
Title: A Phase II Open-label, Single-arm, Multi-center Study of Ruxolitinib Added to Corticosteroids in Pediatric Subjects With Moderate and Severe Chronic Graft vs. Host Disease After Allogeneic Stem Cell Transplantation
Brief Title: Activity, Safety and Pharmacokinetics in Pediatric Subjects With Moderate and Severe Chronic Graft vs. Host Disease After Allogeneic Stem Cell Transplant
Acronym: REACH 5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424G12201; 2018-003296-35 (EudraCT Number)
Record Dates: First submitted 2018-12-11; First posted 2018-12-12 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Graft vs Host Disease
Keywords: GvHD; INC424; pediatric; Chronic Graft versus Host Disease; moderate and severe chronic graft vs. host disease; allogeneic stem cell transplant; ruxolitinib; corticosteroids
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome; Lymphoma, Follicular | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INC424 (ruxolitinib) (Experimental): All pediatric participants received ruxolitinib twice a day (BID) in either tablet or oral solution (liquid), depending on the group they were in.
  Interventions: Drug: INC424

INTERVENTIONS:
Drug: INC424 — Ruxolitinib was taken orally based on age groups as follows:
  Group 1 (>=12y to <18y): 10mg bid as tablet Group 2 (>=6y to <12y): 5mg bid as tablet or liquid Group 3 (>=2y to <6y): 4mg/m2 bid as liquid
  Other Names: Ruxolitinib

SUMMARY:
This open-label, single-arm, Phase II multi-center study enrolled 46 participants and investigated the activity, pharmacokinetics and safety of ruxolitinib added to the subject's immunosuppressive regimen among infants, children, and adolescents aged ≥28 days to <18 years old with either moderate to severe treatment-naive cGvHD or SR-cGvHD.

Although 46 participants were enrolled,1 participant (enrolled in the ≥6y to <12y age group) received study treatment beyond protocol requirements and was excluded from analyses.

DETAILED DESCRIPTION:
Subjects were grouped according to their age as follows:

* Group 1 included subjects ≥12y to <18y
* Group 2 included subjects ≥6y to <12y
* Group 3 included subjects ≥2y to <6y and
* Group 4 included subjects ≥28days to <2y. Enrollment initiation into the youngest age group, Group 4, was subject to the availability of data in this age group from another study, as well as a review of available PK, safety, and activity data generated from Groups 1 to 3 in the current study. At least 5 evaluable participants per group were needed for the primary analysis in Groups 1, 2 and 3. No minimum number of evaluable participants were needed in Group 4. Enrollment was completed prior to the availability of the data and so no subjects were enrolled in Group 4.

After a screening period of Day -28 to Day -1: eligible subjects started study treatment on Cycle

1 Day 1 and were treated for up to a maximum of 3 years (39 cycles/156 weeks) or until early discontinuation. Subjects who discontinued study treatment for any reason earlier than 39 cycles were followed every 6 months until 3 years from their first dose of study treatment was reached.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age ≥28 days and <18 years at the time of informed consent.
* Subjects who have undergone a successful alloSCT from any donor source (matched unrelated donor, sibling, haplo-identical) using bone marrow, peripheral blood stem cells, or cord blood. Recipients of myeloablative or reduced intensity conditioning are eligible.
* Subjects with diagnosed moderate to severe cGvHD according to NIH 2014 Consensus Criteria prior to Cycle 1 Day 1. Other possible diagnoses for clinical symptoms supporting cGvHD diagnoses must be excluded (e.g., infection, drug side effects, malignancy). Subjects must be either:

  * Treatment-naive cGvHD subjects that have not received any prior systemic treatment for cGvHD except for a maximum 72h of prior systemic corticosteroid therapy of methylprednisolone or equivalent after the onset of chronic GvHD. Subjects are allowed to have received prior systemic treatment for cGvHD prophylaxis (as long as the prophylaxis was started prior to the diagnosis of cGvHD).

OR o Steroid-refractory moderate to severe cGvHD as per institutional criteria, or per physician decision in case institutional criteria are not available, and still receiving systemic corticosteroids for the treatment of cGvHD for a duration of <18 months prior to Cycle 1 Day 1. In case the corticosteroids were previously interrupted due to response, the duration of < 18 months applies to the last period of corticosteroid use.

Exclusion Criteria:

* SR-cGvHD subjects with a prior cGvHD treatment with a JAK1- or a JAK2- or a JAK1/2-inhibitor, except when the subject achieved complete or partial response and has been off JAK inhibitor treatment for at least 4 weeks prior to Cycle Day 1 or up to 5 times the half-life of the prior JAK inhibitor, whichever is longer.

  * Subjects who initiated systemic calcineurin inhibitors (CNI; cyclosporine or tacrolimus) within 3 weeks prior to start of ruxolitinib on Cycle 1 Day 1. Note: systemic CNI are allowed when initiated > 3 weeks from start of ruxolitinib.
* Failed prior alloSCT within the past 6 months
* Significant respiratory disease including subjects who are on mechanical ventilation or who have a resting oxygen saturation < 90% by pulse-oximetry on room-air.
* Impairment of gastrointestinal (GI) function (unrelated to GvHD) or GI disease (unrelated to GvHD) that may significantly alter the absorption of oral ruxolitinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection),
* Cholestatic disorders, or unresolved sinusoidal obstructive syndrome/veno-occlusive disease of the liver (defined as persistent bilirubin abnormalities not attributable to cGvHD and ongoing organ dysfunction)
* Presence of clinically active uncontrolled infection including significant bacterial, fungal, viral or parasitic infection requiring treatment.
* Known human immunodeficiency virus (HIV) infection.
* Evidence of uncontrolled hepatitis B virus (HBV) or hepatitis C virus (HCV) based on assessment done by Investigator or delegate.
* Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds.
* History of bone disorders such as osteogenesis imperfecta, rickets, renal osteodystrophy, osteomyelitis, osteopenia, fibrous dysplasia, osteomalacia etc. prior to the underlying diagnosis which resulted in the alloSCT.
* History of endocrine or kidney related growth retardation prior to the underlying diagnosis which resulted in the alloSCT.
* Evidence of clinically active tuberculosis (clinical diagnosis per local practice)
* Any corticosteroid therapy for indications other than cGvHD at doses > 1 mg/kg/daymethylprednisolone (or equivalent prednisone dose 1.25 mg/kg/day) within 7 days of the screening visit.
* History of progressive multifocal leuko-encephalopathy (PML).
* Presence of severely impaired renal function

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2024-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- Novartis Investigative Site, São Paulo, Brazil
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Prague, Czechia
- India (4):
  - Novartis Investigative Site, Tamil Nadu, Chennai
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Bangalore
  - Novartis Investigative Site, Delhi
- Novartis Investigative Site, Roma, RM, Italy
- Japan (2):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Saitama
- Novartis Investigative Site, Saint Petersburg, Russia
- Novartis Investigative Site, Bratislava, Slovakia
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Zurich, Switzerland
- Novartis Investigative Site, Taipei, Taiwan
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Antalya

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Locatelli F, Antmen B, Kang HJ, Koh K, Takahashi Y, Kupesiz A, Dias Matos MGA, Chopra Y, Bhat S, Im HJ, Gungor T, Lu MY, Stefanelli T, Rosko C, St Pierre A, Burock K, Smith Y, Sinclair K, Diaz-de-Heredia C. Ruxolitinib in treatment-naive or corticosteroid-refractory paediatric patients with chronic graft-versus-host disease (REACH5): interim analysis of a single-arm, multicentre, phase 2 study. Lancet Haematol. 2024 Aug;11(8):e580-e592. doi: 10.1016/S2352-3026(24)00174-1. Epub 2024 Jul 10. PMID 39002551
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2541

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At least 5 evaluable participants per group were needed for the primary analysis in Groups 1, 2 and 3. No minimum number of evaluable participants were needed in Group 4.
  Disposition and Demographics are presented by age group.
Pre-assignment Details: Enrollment initiation into the youngest age group, Group 4, was subject to the availability of data in this age group from study CINC424F12201. However, no participants were enrolled in group 4 (aged ≥ 28 days to < 2y) due to the completion of the overall study enrolment with participants in the older age groups (groups 1, 2, & 3).
Groups:
- ≥ 12y - < 18y RUX 10mg BID (Group 1): Participants received ruxolitinib 10mg orally twice a day (BID).
- ≥ 6y - < 12y RUX 5mg BID (Group 2): Participants received ruxolitinib 5mg orally twice a day (BID).
- ≥ 2y - < 6y RUX 4mg/m2 BID (Group 3): Participants received ruxolitinib 4mg/m2 orally twice a day (BID).
Period: Overall Study
Arm/Group | ≥ 12y - < 18y RUX 10mg BID (Group 1) | ≥ 6y - < 12y RUX 5mg BID (Group 2) | ≥ 2y - < 6y RUX 4mg/m2 BID (Group 3)
Started | 22 | 17 | 7
Full Analysis Set (Full Analysis Set comprised all subjects to whom study treatment has been assigned and who received at least one dose of study treatment.) | 22 | 16 | 7
Completed Treatment | 3 | 5 | 3
Discontinued From Treatment | 19 | 11 | 4
Participants Who Received Tablets | 22 | 14 | 0
Participants Who Received Liquid | 0 | 2 | 7
Completed | 14 | 10 | 4
Not Completed | 8 | 7 | 3
Not completed — Death | 6 | 3 | 2
Not completed — Subject decision | 0 | 3 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Guardian decision | 0 | 0 | 1
Not completed — Enrolled but received treatment beyond protocol requirement | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) comprised all subjects to whom study treatment has been assigned and who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | ≥ 12y - < 18y RUX 10mg BID (Group 1) | ≥ 6y - < 12y RUX 5mg BID (Group 2) | ≥ 2y - < 6y RUX 4mg/m2 BID (Group 3) | Total
Number analyzed (Participants) | 22 | 16 | 7 | 45
Age, Continuous [Mean (Standard Deviation); unit: months] | 175.2 (20.05) | 99.3 (18.39) | 47.1 (15.08) | 128.3 (52.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 2 | 16
  Male | 15 | 9 | 5 | 29
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 8 | 10 | 3 | 21
  Black or African American | 0 | 1 | 0 | 1
  Asian | 14 | 5 | 4 | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) at Cycle 7 Day 1
Description: ORR is defined as the percentage of participants demonstrating a complete response (CR) or partial response (PR) without the requirement of additional systemic therapies for an earlier progression, mixed response or non-response. The response is assessed per National Institute of Health (NIH) consensus criteria and scoring of response was relative to the organ stage at the start of study treatment.
Time Frame: At Cycle 7 Day 1 (Day 168); Cycle = 28 Days
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- All Participants: All participants from Group 1, Group 2 and Group 3.
Arm/Group | ≥ 12y - < 18y RUX 10mg BID (Group 1) | ≥ 6y - < 12y RUX 5mg BID (Group 2) | ≥ 2y - < 6y RUX 4mg/m2 BID (Group 3) | All Participants
Number analyzed (Participants) | 22 | 16 | 7 | 45
Percentage of participants | 36.4 [19.6 to 56.1] | 50.0 [27.9 to 72.1] | 28.6 [5.3 to 65.9] | 40.0 [27.7 to 53.3]

2. Secondary Outcome: Ruxolitinib Concentrations by Timepoint
Description: Pharmacokinetics (PK) of ruxolitinib by age groups (and formulation tablet vs liquid).
Time Frame: Cycle 1 Day 1: 0.5, 2 and 6 hours post-dose; Pre-dose on Cycle 1 Day 8, Cycle 1 Day 15, Cycle 1 Day 22, Cycle 3 Day 1, Cycle 5 Day 1 and Cycle 7 Day 1; Cycle = 28 Days
Population: The Pharmacokinetic Analysis Set (PAS) included all subjects who provided at least one evaluable PK concentration. Evaluable PK concentration: Participants took the dose of ruxolitinib prior to PK sample; For post-dose samples on Cycle 1 Day 1: participants did not vomit within 2 hours after dosing with ruxolitinib; For pre-dose samples: participant samples were collected before the next dose administration of ruxolitinib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Groups:
- ≥ 12y - < 18y RUX 10mg BID (Tablet): Participants in this group were administered 10mg ruxolitinib tablet twice a day.
- ≥ 6y - < 12y RUX 5mg BID (Tablet): Participants in this group were administered 5mg ruxolitinib tablets twice a day.
- ≥ 6y - < 12y RUX 5mg BID (Liquid); ≥ 2y - < 6y RUX 4mg/m2 BID (Liquid): Participants in this group were administered ruxolitinib oral pediatric formulation twice a day.
Arm/Group | ≥ 12y - < 18y RUX 10mg BID (Tablet) | ≥ 6y - < 12y RUX 5mg BID (Tablet) | ≥ 6y - < 12y RUX 5mg BID (Liquid) | ≥ 2y - < 6y RUX 4mg/m2 BID (Liquid)
Number analyzed (Participants) | 21 | 13 | 2 | 7
ug/ml
  Cycle 1 Day 1: 0.5 hour (hr) (post-dose): number analyzed (Participants) | 7 | 9 | 1 | 7
  Cycle 1 Day 1: 0.5 hour (hr) (post-dose) | 60.0 (350.7) | 32.4 (471.9) | 78.6 | 60.1 (98.7)
  Cycle 1 Day 1: 2 hr (post-dose): number analyzed (Participants) | 7 | 7 | 1 | 7
  Cycle 1 Day 1: 2 hr (post-dose) | 112 (51.8) | 106 (39.2) | 77.0 | 49.7 (30.7)
  Cycle 1 Day 1: 6hr (post-dose): number analyzed (Participants) | 7 | 8 | 1 | 7
  Cycle 1 Day 1: 6hr (post-dose) | 56.7 (73.9) | 47.8 (164.1) | 60.0 | 15.3 (66.2)
  Cycle 1 Day 8: 0 hr (pre-dose): number analyzed (Participants) | 20 | 13 | 1 | 7
  Cycle 1 Day 8: 0 hr (pre-dose) | 16.7 (208.3) | 10.9 (146.5) | 3.47 | 3.88 (152.4)
  Cycle 1 Day 15: 0 hr (pre-dose): number analyzed (Participants) | 19 | 12 | 2 | 7
  Cycle 1 Day 15: 0 hr (pre-dose) | 17.8 (195.5) | 12.9 (248.2) | 4.14 (399.3) | 9.43 (121.5)
  Cycle 1 Day 22: 0 hr (pre-dose): number analyzed (Participants) | 18 | 11 | 2 | 7
  Cycle 1 Day 22: 0 hr (pre-dose) | 20.8 (199.5) | 11.7 (165.4) | 4.89 (505.2) | 10.3 (150.4)
  Cycle 3 Day 1: 0 hr (pre-dose: number analyzed (Participants) | 17 | 11 | 2 | 5
  Cycle 3 Day 1: 0 hr (pre-dose | 11.4 (193.8) | 11.3 (193.1) | 2.66 (587.5) | 5.56 (180.8)
  Cycle 5 Day 1: 0 hr (pre-dose: number analyzed (Participants) | 14 | 10 | 2 | 4
  Cycle 5 Day 1: 0 hr (pre-dose | 13.0 (176.6) | 16.4 (470.7) | 11.0 (83.5) | 7.32 (102.0)
  Cycle 7 Day 1: 0 hr (pre-dose: number analyzed (Participants) | 12 | 8 | 2 | 4
  Cycle 7 Day 1: 0 hr (pre-dose | 14.3 (173.7) | 10.7 (129.9) | 5.79 (120.1) | 4.94 (165.9)

3. Secondary Outcome: Duration of Response (DOR)
Description: Time from first response until chronic Graft vs. host disease (cGvHD) progression, death, or the date of addition of systemic therapies for cGvHD assessed for responders only based on BOR up to Cycle 7 Day 1. Presented as percentage of participants to still be in response at different time points in months (per Kaplan-Meier estimates). Participants without event will be censored at the date of their last response assessment prior to or at the analysis cut-off date if no events occurred on or before 12 weeks (84 days) after the last GvHD assessment. As planned in the SAP, this outcome measure is provided for all participants instead of per age groups.
Time Frame: From baseline up to 39 cycles; Cycle = 28 Days
Population: FAS comprised all subjects to whom study treatment has been assigned and who received at least one dose of study treatment. Duration of response (DOR) is assessed for responders only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Participants: DOR was analyzed for all responders from the three age groups (Groups 1, 2 and 3)
Arm/Group | All Participants
Number analyzed (Participants) | 37
Percentage of participants
  Month 1 | 94.59 [80.07 to 98.62]
  Month 2 | 86.23 [70.01 to 94.03]
  Month 6 | 74.24 [56.17 to 85.74]
  Month 12 | 63.10 [43.74 to 77.38]
  Month 18 | 58.89 [39.23 to 74.12]
  Month 24 | 58.89 [39.23 to 74.12]
  Month 30 | 58.89 [39.23 to 74.12]
  Month 36 | 58.89 [39.23 to 74.12]

4. Secondary Outcome: Overall Response Rate (ORR) at Cycle 4 Day 1
Description: ORR is defined as the percentage of participants demonstrating a complete response (CR) or partial response (PR) without the requirement of additional systemic therapies for an earlier progression, mixed response or non-response. The response is assessed per National Institute of Health (NIH) consensus criteria and scoring of response will be relative to the organ stage at the start of study treatment at Cycle 4 Day 1.
Time Frame: At Cycle 4 Day 1 (Day 84); Cycle = 28 Days
Population: FAS comprised all subjects to whom study treatment has been assigned and who received at least one dose of study treatment.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | ≥ 12y - < 18y RUX 10mg BID (Group 1) | ≥ 6y - < 12y RUX 5mg BID (Group 2) | ≥ 2y - < 6y RUX 4mg/m2 BID (Group 3) | All Participants
Number analyzed (Participants) | 22 | 16 | 7 | 45
Percentage of participants | 54.5 [35.3 to 72.9] | 62.5 [39.1 to 82.2] | 42.9 [12.9 to 77.5] | 55.6 [42.3 to 68.3]

5. Secondary Outcome: Best Overall Response (BOR)
Description: Percentage of participants who achieved overall response (complete response (CR) or partial response (PR)) at any time point until Cycle 7 Day 1 or the start of additional systemic therapy for chronic GvHD.
Time Frame: Until Cycle 7 Day 1 (Day 168) or the start of additional systemic therapy for cGvHD; Cycle = 28 Days
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | ≥ 12y - < 18y RUX 10mg BID (Group 1) | ≥ 6y - < 12y RUX 5mg BID (Group 2) | ≥ 2y - < 6y RUX 4mg/m2 BID (Group 3) | All Participants
Number analyzed (Participants) | 22 | 16 | 7 | 45
Percentage of participants | 81.8 [63.1 to 93.5] | 81.3 [58.3 to 94.7] | 85.7 [47.9 to 99.3] | 82.2 [70.2 to 90.8]

6. Secondary Outcome: Failure Free Survival (FFS)
Description: Failure-free survival was defined as the time from date of treatment to any of the following events: i) relapse or recurrence of underlying disease or death due to underlying disease, ii) non-relapse mortality, or iii) addition or initiation of another systemic therapy for cGvHD per Kaplan-Meier estimates. As planned in the SAP, this outcome measure is provided for all participants instead of per age groups.
Time Frame: From baseline up to 39 cycles; Cycle = 28 Days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Participants: FFS was analyzed for all participants from the three age groups (Groups 1, 2 and 3)
Arm/Group | All Participants
Number analyzed (Participants) | 45
Percentage of participants
  Month 1 | 91.11 [78.03 to 96.57]
  Month 2 | 84.44 [70.12 to 92.26]
  Month 6 | 68.89 [53.20 to 80.25]
  Month 12 | 64.44 [48.67 to 76.48]
  Month 18 | 57.78 [42.11 to 70.61]
  Month 24 | 57.78 [42.11 to 70.61]
  Month 30 | 57.78 [42.11 to 70.61]
  Month 36 | 57.78 [42.11 to 70.61]

7. Secondary Outcome: Cumulative Incidence of Malignancy Relapse/Recurrence (MR)
Description: MR was defined as the time from date of treatment assignment to the date of hematologic malignancy relapse/recurrence. Calculated for subjects with underlying hematologic malignant disease. The cumulative incidence (CI) of malignancy relapse/recurrence at 1, 2, 6, 12, 18, 24, 30 and 36 months after start of treatment has been reported. As planned in the SAP, this outcome measure is provided for all participants instead of per age groups.
Time Frame: From baseline up to 39 cycles; Cycle = 28 Days
Population: FAS comprised all subjects to whom study treatment has been assigned and who received at least one dose of study treatment, assessed for subjects with malignancy relapse/occurrence only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Participants: MR was analyzed for all participants with underlying hematologic malignant disease from the three age groups (Groups 1, 2 and 3).
Arm/Group | All Participants
Number analyzed (Participants) | 30
Percentage of participants
  Month 1 | 3.33 [0.23 to 14.80]
  Month 2 | 10.00 [2.47 to 23.88]
  Month 6 | 10.00 [2.47 to 23.88]
  Month 12 | 10.00 [2.47 to 23.88]
  Month 18 | 10.00 [2.47 to 23.88]
  Month 24 | 10.00 [2.47 to 23.88]
  Month 30 | 10.00 [2.47 to 23.88]
  Month 36 | 10.00 [2.47 to 23.88]

8. Secondary Outcome: Non-relapse Mortality (NRM)
Description: NRM is defined as the time from date of treatment assignment to date of death not preceded by underlying disease relapse/recurrence calculated for all participants. The cumulative incidence (CI) of non-relapse mortality at 1, 2, 6, 12, 18, 24, 30 and 36 months after start of treatment has been reported. As planned in the SAP, this outcome measure is provided for all participants instead of per age groups.
Time Frame: From baseline up to 39 cycles; Cycle = 28 Days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Participants: NRM was analyzed for all participants from the three age groups (Groups 1, 2 and 3).
Arm/Group | All Participants
Number analyzed (Participants) | 45
Percentage of participants
  Month 1 | 2.22 [0.17 to 10.28]
  Month 2 | 2.22 [0.17 to 10.28]
  Month 6 | 6.67 [1.70 to 16.53]
  Month 12 | 13.33 [5.34 to 25.02]
  Month 18 | 17.78 [8.23 to 30.28]
  Month 24 | 20.07 [9.80 to 32.93]
  Month 30 | 20.07 [9.80 to 32.93]
  Month 36 | 20.07 [9.80 to 32.93]

9. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of treatment assignment to the date of death due to any cause. As planned in the SAP, this outcome measure is provided for all participants instead of per age groups.
Time Frame: From baseline up to 39 cycles; Cycle = 28 Days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: survival probability in percentage
Groups:
- All Participants: OS was analyzed for all participants from the three age groups (Groups 1, 2 and 3).
Arm/Group | All Participants
Number analyzed (Participants) | 45
survival probability in percentage
  Month 1 | 97.78 [85.25 to 99.68]
  Month 2 | 97.78 [85.25 to 99.68]
  Month 6 | 91.06 [77.90 to 96.55]
  Month 12 | 84.23 [69.73 to 92.15]
  Month 18 | 79.67 [64.57 to 88.87]
  Month 24 | 77.33 [61.94 to 87.11]
  Month 30 | 77.33 [61.94 to 87.11]
  Month 36 | 74.91 [59.26 to 85.26]

10. Secondary Outcome: Percentage of Participants With ≥50% Reduction From Baseline in Daily Corticosteroid Dose
Description: Reduction of at least ≥50% from baseline in daily corticosteroid use by Cycle 7 Day 1 (regardless of reason). As planned in the SAP, this outcome measure is provided for all participants instead of per age groups, for those who received corticosteroids at baseline.
Time Frame: Baseline to Cycle 7 Day 1 (Day 168); Cycle = 28 Days
Population: FAS comprised all subjects to whom study treatment has been assigned and who received at least one dose of study treatment and received corticosteroids at baseline.
Measure: Number; unit: Percentage of participants
Groups:
- All Participants: The percentage of participants with ≥50% reduction from baseline in daily corticosteroid dose at least once was analyzed for all participants in Groups 1, 2 and 3 who received corticosteroids at baseline.
Arm/Group | All Participants
Number analyzed (Participants) | 40
Percentage of participants | 75.0

11. Secondary Outcome: Percentage of Participants With a Reduction to a Low Dose Corticosteriod
Description: Reduction to low dose corticosteroids, is defined as the percentage of participants with reduction from baseline in daily corticosteroid dose to methylprednisolone-equivalent steroid dose of ≤ 0.2 mg/kg/day (or equivalent dose of ≤ 0.25 mg/kg/day prednisone or prednisolone). As planned in the SAP, this outcome measure is provided for all participants instead of per age groups, for those who received corticosteroids at baseline.
Time Frame: Baseline to Cycle 7 Day 1 (Day 168); Cycle = 28 Days
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Groups:
- All Participants: The percentage of participants with reduction to <=0.2mg/kg/day from baseline in daily corticosteroid dose at least once was analyzed for all participants in Groups 1, 2 and 3 who received corticosteroids at baseline.
Arm/Group | All Participants
Number analyzed (Participants) | 40
Percentage of participants | 67.5

12. Secondary Outcome: Graft Failure
Description: Reported are the number of participants with graft failure from all age groups together. Graft failure was assessed by donor cell chimerism, defined as initial whole blood or marrow donor chimerism for those who had ≥ 5% donor cell chimerism at baseline. If donor cell chimerism declined to < 5% on subsequent measurements, graft failure was declared. As planned in the SAP, this outcome measure is provided for all participants instead of per age groups.
Time Frame: From baseline up to 39 cycles; Cycle = 28 Days
Population: FAS comprised all subjects to whom study treatment has been assigned and who received at least one dose of study treatment. As planned in the SAP, this outcome measure is provided for all participants instead of per age groups.
Measure: Number; unit: Participants
Groups:
- All Participants: Graft Failure was analyzed for all participants from the three age groups (Groups 1, 2 and 3).
Arm/Group | All Participants
Number analyzed (Participants) | 45
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and on-treatment deaths were collected from the first dose of study treatment up to 30 days after last dose of study medication. Post-treatment survival follow-up deaths were collected 31 days after last dose of study medication until the end of the study, up to approx. 36 months/39 cycles.
Description: An Adverse Event (AE) is any sign or symptom that occurs during the conduct of the trial and post-treatment survival follow-up.
Groups:
- On-Treatment >=12y - <18y RUX 10mg BID; On-Treatment >=6y - <12y RUX 5mg BID; On-Treatment >=2y - <6y RUX 4mg/m2 BID: On-treatment period: from first dose of study treatment up to 30 days post-treatment.
- On-Treatment - All Participants; Post-Treatment All Participants: All participants from Group 1, Group 2 and Group 3.
- Post-Treatment >=12y - <18y RUX 10mg BID; Post-Treatment >=6y - <12y RUX 5mg BID; Post-Treatment >=2y - <6y RUX 4mg/m2 BID: Events collected in the post- treatment survival follow-up phase (starting from day 31 post- treatment).
Arm/Group | On-Treatment >=12y - <18y RUX 10mg BID | On-Treatment >=6y - <12y RUX 5mg BID | On-Treatment >=2y - <6y RUX 4mg/m2 BID | On-Treatment - All Participants | Post-Treatment >=12y - <18y RUX 10mg BID | Post-Treatment >=6y - <12y RUX 5mg BID | Post-Treatment >=2y - <6y RUX 4mg/m2 BID | Post-Treatment All Participants
All-Cause Mortality (participants affected / at risk) | 0/22 | 2/16 | 1/7 | 3/45 | 6/22 | 1/16 | 1/7 | 8/45
Serious Adverse Events (participants affected / at risk) | 15/22 | 7/16 | 4/7 | 26/45 | 3/22 | 0/16 | 0/7 | 3/45
Other Adverse Events (participants affected / at risk) | 22/22 | 15/16 | 7/7 | 44/45 | 4/22 | 2/16 | 0/7 | 6/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | On-Treatment >=12y - <18y RUX 10mg BID (N=22) | On-Treatment >=6y - <12y RUX 5mg BID (N=16) | On-Treatment >=2y - <6y RUX 4mg/m2 BID (N=7) | On-Treatment - All Participants (N=45) | Post-Treatment >=12y - <18y RUX 10mg BID (N=22) | Post-Treatment >=6y - <12y RUX 5mg BID (N=16) | Post-Treatment >=2y - <6y RUX 4mg/m2 BID (N=7) | Post-Treatment All Participants (N=45)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Human bocavirus infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Transplant failure (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aura (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | On-Treatment >=12y - <18y RUX 10mg BID (N=22) | On-Treatment >=6y - <12y RUX 5mg BID (N=16) | On-Treatment >=2y - <6y RUX 4mg/m2 BID (N=7) | On-Treatment - All Participants (N=45) | Post-Treatment >=12y - <18y RUX 10mg BID (N=22) | Post-Treatment >=6y - <12y RUX 5mg BID (N=16) | Post-Treatment >=2y - <6y RUX 4mg/m2 BID (N=7) | Post-Treatment All Participants (N=45)
Anaemia (Blood and lymphatic system disorders) | 7 | 2 | 2 | 11 | 0 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 2 | 8 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 5 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 3 | 1 | 0 | 4 | 0 | 0 | 0 | 0
Ear canal stenosis (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Astigmatism (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 2 | 1 | 1 | 4 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 4 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1 | 5 | 0 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 0 | 5 | 1 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pain (General disorders) | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 4 | 0 | 7 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Allergy to chemicals (Immune system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
BK virus infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 4 | 3 | 2 | 9 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 2 | 1 | 4 | 0 | 0 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 2 | 2 | 0 | 4 | 0 | 0 | 0 | 0
Epstein-Barr viraemia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 2 | 1 | 4 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 1 | 5 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Oral viral infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 2 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 1 | 0 | 5 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 4 | 9 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Extraskeletal ossification (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1 | 1 | 5 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Blood magnesium increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Epstein-Barr virus test positive (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Herpes simplex test positive (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Immunoglobulins decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 5 | 2 | 2 | 9 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 5 | 2 | 0 | 7 | 1 | 0 | 0 | 1
Serum ferritin increased (Investigations) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Vascular access device culture positive (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 2 | 1 | 5 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 3 | 1 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 4 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypozincaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 3 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 4 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 2 | 0 | 7 | 1 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Acquired phimosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 6 | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 4 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 3 | 1 | 7 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT03774082/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT03774082/SAP_001.pdf